CLINICAL TRIAL: NCT00279331
Title: Implementation of a Third Generation Sentinel Surveillance Approach Among Men Who Have Sex With Men at High Risk for HIV, Type-1 Acquisition in the Andean Region
Brief Title: Estimating the Incidence of HIV Infection Among Men Who Have Sex With Men in Peru and Ecuador
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Comprehensive International Program of Research on AIDS (Other)
Responsible Party: Sponsor
Other Study IDs: CIPRA PE 002; I-U19-AI053218-01A2; Project 3B; 10408 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2006-01-18; First posted 2006-01-19 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: HIV Infections; Syphilis; Sexually Transmitted Diseases
Keywords: HIV Seronegativity; Men who have Sex with Men; MSM; Peru; Ecuador; Incidence; Prevalence; Drug resistance, viral
MeSH Terms: conditions — HIV Infections; Syphilis; Sexually Transmitted Diseases; Homosexuality

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this observational study is to estimate the number of new HIV infections and the number and variability of antiretroviral-resistant HIV strains among men who have sex with men (MSM). Participants will be recruited from four sites in Peru and one site in Ecuador.

DETAILED DESCRIPTION:
The governments of Peru and Ecuador signed an agreement with the Global Fund to Fight AIDS, Tuberculosis, and Malaria to help guarantee comprehensive quality of care to people living with HIV, including access to antiretrovirals (ARVs). Current methods of surveillance are inadequate in estimating the true burden of disease. Broad access to ARVs in countries without regular drug resistance testing can also cause rapid development of ARV resistance. By establishing a more sophisticated surveillance system able to capture HIV incidence, prevalence, patterns of HIV resistance, and genetic variability of viral strains, Peru and Ecuador will be better equipped to monitor the HIV epidemic, develop personalized prevention and control measures, and track patterns of HIV resistance among infected patients. This study will estimate the incidence of HIV, syphilis, and herpes simplex virus 2 (HSV-2) among MSM in Peru and Ecuador, as well as examine the number and variability of ARV-resistant HIV strains.

This study will last about 2 weeks. Medical history, a physical exam, an HIV rapid test, and HIV pre- and post-test counseling will occur at study entry. Those who test HIV positive will be asked to return to the test site in about 2 weeks to receive confirmatory test results. Patients confirmed to be infected with HIV will be referred to HIV treatment clinics in their area.

At study entry, participants will also undergo a syphilis test. Those who test positive for syphilis will receive same-day treatment at the clinic and be asked to return during Week 1 and 2 to complete treatment for sexually transmitted diseases (STDs) according to local guidelines. STD treatment will not be provided by the study. Those who test negative to both the HIV rapid test and the syphilis test at screening will not participate in any more study visits. Patients who consent to having samples stored for further investigations will also have their samples tested for HSV-2 infection following completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* HIV uninfected or unaware of HIV infection status
* Male at birth
* Report having anal intercourse, either insertive or receptive, with another man 6 months prior to study entry
* Living in one of the participating study cities at time of study entry
* Self-report at least one of the following behaviors:

  * No condom use during the last receptive or insertive anal intercourse
  * Receptive or insertive anal intercourse with more than five sex partners 6 months prior to study entry
  * Exchange of money, gifts, drugs, or shelter for sex 6 months prior to study entry
  * STD symptoms 6 months prior to study entry
  * Inconsistent condom use with an HIV infected sex partner 6 months prior to study entry

Exclusion Criteria:

* HIV infected
* Unwilling to participate in HIV screening
* Any psychiatric or mental condition that may interfere with the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2608 (Estimated)
Dates: Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan Guanira, MD, MPH, Study Chair — Asociación Civil Impacta Salud y Educación, Lima, Peru; Jorge Sanchez, MD, MPH, Principal Investigator — Asociación Civil Impacta Salud y Educación, Lima, Peru; Javier R. Lama, MD, MPH, Principal Investigator — Asociación Civil Impacta Salud y Educación, Lima, Peru
Locations (6):
- Fundación Ecuatoriana Equidad CIPRA CRS, Guayaquil-Guayas, Ecuador
- Peru (5):
  - IMPACTA - Miraflores CIPRA CRS, Lima
  - IMPACTA - Lince CIPRA CRS, Lima
  - IMPACTA - San Miguel CIPRA Project 3B CRS, Lima
  - Policlinico Daniel Alcides Carrión CIPRA CRS, Lima
  - Asoc. de Servicios Generales de Salud y Educación CIPRA CRS, Sullana

REFERENCES:
- [Background] Bautista CT, Sanchez JL, Montano SM, Laguna-Torres VA, Lama JR, Sanchez JL, Kusunoki L, Manrique H, Acosta J, Montoya O, Tambare AM, Avila MM, Vinoles J, Aguayo N, Olson JG, Carr JK. Seroprevalence of and risk factors for HIV-1 infection among South American men who have sex with men. Sex Transm Infect. 2004 Dec;80(6):498-504. doi: 10.1136/sti.2004.013094. PMID 15572623
- [Background] Caceres CF, Mendoza W. Monitoring trends in sexual behaviour and HIV/STIs in Peru: are available data sufficient? Sex Transm Infect. 2004 Dec;80 Suppl 2(Suppl 2):ii80-4. doi: 10.1136/sti.2004.012021. PMID 15572646
- [Background] Goodreau SM, Goicochea LP, Sanchez J. Sexual role and transmission of HIV Type 1 among men who have sex with men, in Peru. J Infect Dis. 2005 Feb 1;191 Suppl 1(0 1):S147-58. doi: 10.1086/425268. PMID 15627225
- [Background] Hirsch MS, Brun-Vezinet F, Clotet B, Conway B, Kuritzkes DR, D'Aquila RT, Demeter LM, Hammer SM, Johnson VA, Loveday C, Mellors JW, Jacobsen DM, Richman DD. Antiretroviral drug resistance testing in adults infected with human immunodeficiency virus type 1: 2003 recommendations of an International AIDS Society-USA Panel. Clin Infect Dis. 2003 Jul 1;37(1):113-28. doi: 10.1086/375597. Epub 2003 Jun 23. PMID 12830416